CLINICAL TRIAL: NCT00462865
Title: A Phase II Study of Adjuvant Gemcitabine/Capecitabine and Bevacizumab for Patients Treated Neoadjuvantly Chemotherapy for Early Stage Breast Cancer With High Risk for Relapse
Brief Title: Trial of Chemotherapy and Avastin as Treatment for Women With Breast Cancer at High Risk for Relapse
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: DSMB determined toxicity of regimen more than originally thought. Slow accrual.
Sponsor: Brown University (Other)
Collaborators: Women and Infants Hospital of Rhode Island (Other); Rhode Island Hospital (Other); The Miriam Hospital (Other); Memorial Hospital of Rhode Island (Other); University of New Mexico Cancer Center (Other)
Responsible Party: Principal Investigator, Bachir Sakr, Principal Investigator, Brown University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG BR-213; AVF4173s (Other: Genentech)
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Results first posted 2015-04-08 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
Keywords: breast cancer; neoadjuvant chemotherapy; adjuvant treatment; consolidation therapy; anti-angiogenesis therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine and Capecitabine and Avastin (Experimental): Avastin administered concurrently with chemotherapy (Gemcitabine + Capecitabine) for six cycles followed by single agent Avastin to complete one year of treatment. Radiation therapy (if planned) will take place after adjuvant chemotherapy completes.
  Interventions: Drug: Gemcitabine and Capecitabine and Avastin

INTERVENTIONS:
Drug: Gemcitabine and Capecitabine and Avastin — avastin administered concurrently with chemotherapy (gemcitabine + capecitabine) for six cycles followed by single agent avastin to complete one year of treatment. Radiation therapy (if planned) will take place after adjuvant chemotherapy completes.
  Other Names: Gemzar, Xeloda, Bevacizumab

SUMMARY:
Women with breast cancer who are not eligible for breast conserving surgery or who have node-involvement are sometimes treated with chemotherapy up front, in hopes of allowing for a woman to keep her breast and decreasing the size of the excision for her breast cancer. While current research has shown that survival is the same whether women are treated with chemotherapy first or surgery first for breast cancer, the investigators do not yet know how to treat women with persistent breast cancer after she has received primary chemotherapy. This study looks at the use of a combination regimen of two agents (gemcitabine and capecitabine), both of which are active in breast cancer, and using Avastin to see if this regimen can be given to women treated with primary chemotherapy and then surgery, considered to be at high risk of relapse.

DETAILED DESCRIPTION:
For patients with locally advanced breast cancers (LABC) primary or neoadjuvant chemotherapy (NAC) has become accepted as standard treatment. Advantages of NAC include shrinking the primary tumor, often rendering an unresectable cancer resectable, and the theoretically concurrent treatment of occult metastatic disease prior to definitive local therapy (surgery +/- radiation therapy). NAC can reduce the extent of surgery required for the management of local breast cancer from mastectomy to lump- or segmentectomy, without compromising major outcome measures, such as overall and disease free survival. At this time, the current standard of care for women felt to be candidates for NAC is an anthracycline + taxane regimen. The intent is to induce a pCR which as noted above is a strong indicator of survival. Yet, in both large NSABP studies, the proportion of women achieving this is less than 20% with these regimens raising a major challenge in clinical practice: what is the appropriate treatment for women with persistent disease after NAC? Given that gemcitabine and capecitabine are non-cross-resistant to anthracyclines and taxanes and use a different mechanism of action, have an acceptable toxicity profile, and in the absence of standard options for therapy we are interested in utilizing these agents coupled with bevacizumab as adjuvant treatment in women with residual breast cancer following primary chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

General health

* Women Age >18.
* ECOG Performance status 0-1
* Life expectancy must be 3 months. Clinical stage
* Histologically or cytologically adenocarcinoma of breast
* Pre-operative stage II-III per AJCC 6th edition, based on baseline evaluation by clinical examination, breast imaging, and/or preoperative work-up.
* Evidence of residual invasive breast cancer or node positive disease following neoadjuvant chemotherapy.

Prior Therapy

* Patients must have received primary (neoadjuvant) chemotherapy for local or locoregional breast cancer containing an anthracycline and a taxane.
* Patients must have completed definitive resection of primary tumor with adequate excision of gross disease.
* Patients must have residual invasive carcinoma in the breast and/or residual carcinoma in one or more regional nodes following preoperative chemotherapy.

Adequate hematologic and metabolic parameters within four weeks of study entry defined as:

* Absolute neutrophil count ≥1,500/mm3 Platelets ≥ 150,000/mm3
* Total bilirubin ≤ 2.0 mg/dL
* Serum creatinine ≤ 2x upper limit of normal
* Serum calcium ≤1.5x upper normal limit Concurrent treatments
* Current use of anti-coagulants is allowed as long as patients have been on a stable dose for more than 2 weeks with stable INR.
* Chronic therapy with full dose aspirin up to 325 mg/day or standard non-steroidal anti-inflammatory agents is allowed.

Informed consent

* Provision of signed informed consent.

Exclusion Criteria:

Prior therapy

* No prior gemcitabine, continuous infusion 5-FU, or oral fluoropyrimidine (capecitabine, UFT, S-1, 5-FU/eniluracil, etc.)
* No known hypersensitivity to capecitabine or prior unanticipated severe reaction to (capecitabine, UFT, S-1, 5-FU/eniluracil, etc.) therapy or known hypersensitivity to 5-fluorouracil.
* No concurrent or prior endocrine therapy as adjuvant treatment.
* No prior breast radiation
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in another experimental drug study
* Stage IV breast cancer
* Patients must not have evidence of metastatic disease at enrollment. Women of child-bearing potential.
* Nonpregnant and nonlactating.
* Women of child-bearing potential must have a negative serum pregnancy test and must agree to an effective means of contraception during the entire study period.

Concurrent medical conditions:

* No other active cancers, except non-melanoma skin cancers.
* No serious infection or other serious underlying medical condition that would otherwise impair their ability to receive protocol treatment.
* Patients with clinically significant medical or psychiatric problems which may interfere with treatment on study.

Avastin-specific exclusions:

* Inadequately controlled hypertension (defined as systolic blood pressure 150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* Known CNS disease
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Serious, non-healing wound, ulcer, or bone fracture
* Proteinuria at screening as demonstrated by urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour
* urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).
* Known hypersensitivity to any component of bevacizumab any history of stroke or transient ischemic attack at any time
* History of myocardial infarction or unstable angina within 12 months of study enrollment Inability to comply with study and/or follow-up procedures

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-11; Primary Completion 2012-03 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bachir Sakr, MD, Principal Investigator — Women & Infants' Hospital of Rhode Island; William Sikov, MD, Principal Investigator — Lifespan Hospitals; Melanie Royce, MD, Principal Investigator — University of New Mexico Cancer Center
Locations (3):
- United States (3):
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Lifespan Hospitals, Providence, Rhode Island
  - Women & Infants' Hospital, Providence, Rhode Island

REFERENCES:
- [Background] Sikov WM, Theall KP, Seidler CW, Strenger RS, Fenton MA. Gemcitabine and capecitabine in metastatic breast cancer (MBC): A Brown University Oncology Group (BrUOG) Proc ASCO; 2005; Orlando, FL; 2005. p. 785.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 women enrolled from 3 hospitals, 17 treated
Groups:
- Gemcitabine, Capectiabine, Avastin: After completion of neoadjuvant as well as surgical therapy the combination of gemcitabine/ Capecitabine and Avastin will be given for a total of six cycles.
  Doses to be administered:
  Gemcitabine 2000 mg/m2 on D1 Capecitabine 650 mg/m2 BID on D1-14 Avastin 15 mg/kg on D1
  Following six cycles, patients will proceed to comprehensive breast radiation (if indicated) and will continue to receive avastin every 3 weeks during and after radiotherapy to complete 1 year of treatment.
Period: Overall Study
Arm/Group | Gemcitabine, Capectiabine, Avastin
Started | 18 (18 pts enrolled,1 pt experienced a SAE infection normal ANC (gr 3) and did not begin study,see SAE)
Completed | 17
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment: After completion of neoadjuvant as well as surgical therapy the combination of gemcitabine/ Capecitabine and Avastin will be given for a total of six cycles.
  Doses to be administered:
  Gemcitabine 2000 mg/m2 on D1 Capecitabine 650 mg/m2 BID on D1-14 Avastin 15 mg/kg on D1
  Following six cycles, patients will proceed to comprehensive breast radiation (if indicated) and will continue to receive avastin every 3 weeks during and after radiotherapy to complete 1 year of treatment.
Arm/Group | Treatment
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Toxicity Related to Treatment
Description: 6 out of 17 patients came off study for toxicity prior to receiving all treatment. Toxicity issues of administering 6 cycles of gemcitabine, capecitabine, and Avastin and one year of consolidation of Avastin in women with breast cancer previously treated with neoadjuvant chemotherapy that lead to patients being taken off study.
Time Frame: 1 year
Measure: Number; unit: participants
Groups:
- Gemcitabine, Capectiabine, Avastin: After completion of neoadjuvant as well as surgical therapy the combination of gemcitabine/ Capecitabine and Avastin will be given for a total of six cycles that lead to patients being taken off study.
  Doses to be administered:
  Gemcitabine 2000 mg/m2 on D1 Capecitabine 650 mg/m2 BID on D1-14 Avastin 15 mg/kg on D1
  Following six cycles, patients will proceed to comprehensive breast radiation (if indicated) and will continue to receive avastin every 3 weeks during and after radiotherapy to complete 1 year of treatment.
Arm/Group | Gemcitabine, Capectiabine, Avastin
Number analyzed (Participants) | 17
participants | 6

2. Secondary Outcome: Number of Participants With Recurrent Disease
Time Frame: 6 months and again at the end of the study (1 year)
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine, Capectiabine, Avastin
Number analyzed (Participants) | 18
Participants | 4

ADVERSE EVENTS:
Time Frame: every 3 cycles then off study, for up to 1.5 years (once off study)
Arm/Group | Gemcitabine, Capectiabine, Avastin
Serious Adverse Events (participants affected / at risk) | 5/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Capectiabine, Avastin (N=17)
Left ventricular dysfunction (3) (Investigations) | 1 (1)
infection normal ANC (3) (Investigations) | 2 (2)
pneumonia (3) (Investigations) | 1 (1)
anxiety, distress, diarrhea, headache, dehydration, dizziness, bilateral SOB (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Capectiabine, Avastin (N=17)
abdominal distress/pain (Investigations) | 2 (2)
agitation (Investigations) | 1 (1)
Albumin (Investigations) | 1 (1)
Alk Phos (Investigations) | 5 (5)
alopecia (Investigations) | 2 (2)
ALT (Investigations) | 9 (9)
ANC (Investigations) | 1 (1)
anemia (Investigations) | 1 (1)
anorexia (Investigations) | 3 (3)
anxiety/panic attack (Investigations) | 2 (2)
arthraglias (Investigations) | 1 (1)
AST (Investigations) | 10 (10)
Bili (Investigations) | 2 (2)
bleeding gums (Investigations) | 1 (1)
bloat (Investigations) | 1 (1)
bradycardia (Investigations) | 1 (1)
CA (Investigations) | 2 (2)
constipation (Investigations) | 6 (6)
cough (Investigations) | 2 (2)
Creatinine (Investigations) | 2 (2)
dehydration (Investigations) | 2 (2)
diabetic issue (Investigations) | 1 (1)
diarrhea (Investigations) | 4 (4)
dizziness (Investigations) | 1 (1)
dry skin (Investigations) | 1 (1)
DVT (Investigations) | 1 (1)
dysgeuisa (Investigations) | 4 (4)
dysphagia (Investigations) | 1 (1)
edema (Investigations) | 5 (5)
epistaxis (Investigations) | 1 (1)
erythema (Investigations) | 2 (2)
esophagitis (Investigations) | 1 (1)
fatigue (Investigations) | 12 (12)
fibromyalgia (Investigations) | 1 (1)
genital lesion (Investigations) | 1 (1)
GI other (Investigations) | 2 (2)
Glucose (Investigations) | 2 (2)
hand and foot (Investigations) | 7 (7)
hemmarhoids (Investigations) | 1 (1)
Hgb (Investigations) | 4 (4)
hoarseness (Investigations) | 1 (1)
hot flash (Investigations) | 2 (2)
HTN (Investigations) | 7 (7)
hyperbilrubemia (Investigations) | 1 (1)
hyperglycemia (Investigations) | 1 (1)
hyperpigmentation (Investigations) | 2 (2)
Hyponatremia (Investigations) | 1 (1)
hypotension (Investigations) | 1 (1)
infection normal ANC (Investigations) | 4 (4)
insomnia (Investigations) | 2 (2)
K (Investigations) | 2 (2)
LDH (Investigations) | 1 (1)
left nostril pain (Investigations) | 1 (1)
left ventricular dysfunction (Investigations) | 1 (1)
LFTs (Investigations) | 1 (1)
loss of vision (Investigations) | 1 (1)
Mg (Investigations) | 6 (6)
mood alteration (Investigations) | 1 (1)
mouth sores (Investigations) | 1 (1)
mucositis (Investigations) | 4 (4)
muscle cramps (Investigations) | 1 (1)
nasal dryness (Investigations) | 1 (1)
nausea (Investigations) | 7 (7)
neuropathy (Investigations) | 6 (6)
pain- muscosk (Investigations) | 14 (14)
pharyngitis (Investigations) | 2 (2)
Phos (Investigations) | 2 (2)
Plts (Investigations) | 3 (3)
proteinuria (Investigations) | 1 (1)
pruritis (Investigations) | 1 (1)
rash (Investigations) | 3 (3)
rectal bleed/pain (Investigations) | 3 (3)
rhinitis (Investigations) | 2 (2)
rigor (Investigations) | 1 (1)
scalp blisters (Investigations) | 1 (1)
sinusitis (Investigations) | 1 (1)
SOB (Investigations) | 2 (2)
somolence (Investigations) | 1 (1)
tachycardia (Investigations) | 1 (1)
thrombocytopenia (Investigations) | 1 (1)
tremor (Investigations) | 1 (1)
Uric Acid (Investigations) | 1 (1)
Urine Protein (Investigations) | 1 (1)
vaginitis (Investigations) | 1 (1)
vomitting (Investigations) | 5 (5)
WBC (Investigations) | 5 (5)
wound healing delay (Investigations) | 1 (1)
wt loss (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No